CLINICAL TRIAL: NCT03300635
Title: Metaboliset Muutokset ja Lihastoiminta Fibromyalgiassa
Brief Title: Metabolism, Muscle Function and Psychological Factors in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Ritva Markkula, Principal Investigator, specialist doctor, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TYH2017215
Record Dates: First submitted 2017-09-12; First posted 2017-10-03 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Glucose Tolerance Test; Exercise Test

STUDY DESIGN:
Intervention Model Description: Patients and healthy control subjects will attend the same interventions: a) muscle function test (distressing task vs. relaxing) with e.g. psychological questionnaires, b) glucose tolerance test and other blood analyses including metabolomics, and c) bicycle ergometry with physiological measurements and blood analyses including metabolomics.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibromyalgia patients (Other): All study subjects, both patients and healthy controls, will attend all three interventions: Mental distress and relaxation test, Glucose tolerance test, and Exercise test
  Interventions: Other: Mental distress and relaxation test; Other: Glucose tolerance test; Other: Exercise test
- Healthy controls (Other): All study subjects, both patients and healthy controls, will attend all three interventions: Mental distress and relaxation test, Glucose tolerance test, and Exercise test
  Interventions: Other: Mental distress and relaxation test; Other: Glucose tolerance test; Other: Exercise test

INTERVENTIONS:
Other: Mental distress and relaxation test
Other: Glucose tolerance test
Other: Exercise test

SUMMARY:
Fibromyalgia (FM) is a world widely common syndrome, characterized by widespread pain, often accompanied by general fatigue, soreness, and abnormal sensations (like "pins and needles"). The reasons and the mechanisms (pathogenesis) of FM are still poorly understood. Efficacious therapies cannot be developed without understanding the pathophysiological mechanisms of the disease or syndrome.

FM patients suffer from pain and sense of weakness and fatigue in the muscles, and often report difficulty in relaxing their muscles. So far, the studies on muscle activation in fibromyalgia (mostly using surface electromyography) have shown some unusual functioning, a kind of overuse, but the results have been somewhat contradictory.

FM symptoms share some features with small fibre neuropathy, which is a disease or abnormality of small nerve fibres with a diverse aetiology. Recently, several research groups have shown (studying both the electrical function of superficial nerves and nerve endings of skin samples) that up to 50% of the FM patients with severe symptoms have small fibre neuropathy: their small nerves do not function properly and small nerve fibre density in their skin is reduced. However, as this phenomenon is common but not a rule, it might be rather a consequence of some underlying mechanisms of the syndrome, creating even more symptoms.

The aim is to investigate whether there would exist metabolic changes in FM patients that would create pain and lead to functional changes and damage in small nerve fibres. The investigators also aim to explore the muscle function particularly in distressed situations and at rest. The hypothesis is that a towards-overuse-altered function would create unfavourable metabolic changes. Third, the aim is to investigate some psychological factors (such as tendency to get anxious or distressed) to find out, if there is any association between them and muscle function.

The FM patients as well as healthy control subjects will be recruited at Helsinki University Hospital Pain Clinic and from primary care at Vantaa Health Care Centre. The voluntary test subjects will attend

1. A muscle function examination of 30 minutes with electromyography using surface electrodes, including mentally distressing tasks and relaxing periods. At the same session, the subject will reply to some questionnaires regarding their symptoms and measuring some psychological factors. Actual pain level will be assessed.
2. A glucose tolerance test, with other blood samples
3. A bicycle ergometer exercise test of 20 - 30 minutes, with both physiological and chemical (blood samples) recordings. Actual pain level will be assessed as well.

At this stage, 40 patients and 20 healthy control subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* fibromyalgia diagnosed by the researchers RM or TZ, based on the ACR criteria from 1990
* Finnish as native language

Exclusion Criteria:

* male sex
* muscular or neuromuscular diseases
* diabetes
* heart disease
* generalised atherosclerosis
* untreated hypertension
* neurological or other disease that systematically affects muscles
* a severe psychiatric disorder
* regular consumption of beta-blockers, bronchodilators, or statins

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The Finnish personal ID system includes identification of gender. As most of clinical FM patients are women, we exclude men to create as much homogenity as possible in our sample.
Enrollment: 81 (Actual)
Dates: Start 2015-09-05 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
metabolomics | up to day 3
  the difference of value distribution in metabolics panel between groups
metabolomics (physical stress) | Day 3 (at the end of Exercise test)
  the difference of value distribution in metabolics panel between groups
metabolomics (metabolic stress) | Day 2 ( at the end of Glucose test)
  the difference of value distribution in metabolics panel between groups
muscle function (raw) | Day 1
  sEMG signal amplitude
muscle function (normalized) | Day 1
  normalized signal amplitude (%sEMGmax)
muscle rest time | Day 1
  time of sEMG signal amplitude < 0.5% sEMGmax

SECONDARY OUTCOMES:
Perceived distress during mental stress vs. relaxation (baseline) | Day 1 ( at the beginning of the recording during the Mental distress and relaxation test)
  reported distress intensity (NRS)
Perceived distress during mental stress vs. relaxation (relaxation I) | Day 1 (after the first relaxation phase of the Mental distress and relaxation test)
  reported distress intensity (NRS)
Perceived distress during mental stress vs. relaxation (mental stress I) | Day 1 (after the first mental stress phase of the Mental distress and relaxation test)
  reported distress intensity (NRS)
Perceived distress during mental stress vs. relaxation (relaxation II) | Day 1 (after the second relaxation phase of the Mental distress and relaxation test)
  reported distress intensity (NRS)
Perceived distress during mental stress vs. relaxation (mental stress II) | Day 1 (after the second mental stress phase of the Mental distress and relaxation test)
  reported distress intensity (NRS)
Perceived distress during mental stress vs. relaxation (relaxation III) | Day 1 ( after the third relaxation phase of the Mental distress and relaxation test)
  reported distress intensity (NRS)
Pain intensity during mental stress vs. relaxation (baseline) | Day 1 ( at the beginning of the recording during the Mental distress and relaxation test)
  reported pain intensity (NRS)
Pain intensity during mental stress vs. relaxation (relaxation I) | Day 1 ( after the first relaxation phase of the Mental distress and relaxation test)
  reported pain intensity (NRS)
Pain intensity during mental stress vs. relaxation (mental stress I) | Day 1 ( after the first mental stress phase of the Mental distress and relaxation test)
  reported pain intensity (NRS)
Pain intensity during mental stress vs. relaxation (relaxation II) | Day 1 (after the second relaxation phase of the Mental distress and relaxation test)
  reported pain intensity (NRS)
Pain intensity during mental stress vs. relaxation (mental stress II) | Day 1 (after the second mental stress phase of the Mental distress and relaxation test)
  reported pain intensity (NRS)
Pain intensity during mental stress vs. relaxation (relaxation III) | Day 1 (after the third relaxation phase of the Mental distress and relaxation test)
  reported pain intensity (NRS)
heart rate variability | Day 1
  variability of heart beat interval evaluated as root mean square successive difference (RMSSD)

CONTACTS AND LOCATIONS:
Overall Officials: Eija A Kalso, MD, PhD, Study Chair — Helsinki University Hospital and Helsinki University
Locations (1):
- HelsinkiUCH, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available for only two of the researchers, Ritva Markkula and Teemu Zetterman, who are recruiting the subjects and collecting and coding their personal data to an unidentified mode.

REFERENCES:
- [Derived] Lehto T, Zetterman T, Gagnon D, Markkula R, Arokoski J, Kalso E, Peltonen JE. Muscle and cerebral oxygenation during exercise in fibromyalgia: a near-infrared spectroscopy study. Eur J Appl Physiol. 2025 Oct 9. doi: 10.1007/s00421-025-06013-8. Online ahead of print. PMID 41065862
- [Derived] Lehto T, Zetterman T, Markkula R, Arokoski J, Tikkanen H, Kalso E, Peltonen JE. Cardiac output and arteriovenous oxygen difference contribute to lower peak oxygen uptake in patients with fibromyalgia. BMC Musculoskelet Disord. 2023 Jul 1;24(1):541. doi: 10.1186/s12891-023-06589-2. PMID 37393269
- [Derived] Zetterman T, Markkula R, Miettinen T, Kalso E. Heart rate variability responses to cognitive stress in fibromyalgia are characterised by inadequate autonomous system stress responses: a clinical trial. Sci Rep. 2023 Jan 13;13(1):700. doi: 10.1038/s41598-023-27581-9. PMID 36639565
- [Derived] Zetterman T, Markkula R, Kalso E. Elevated highly sensitive C-reactive protein in fibromyalgia associates with symptom severity. Rheumatol Adv Pract. 2022 Jun 25;6(2):rkac053. doi: 10.1093/rap/rkac053. eCollection 2022. PMID 35832286
- [Derived] Zetterman T, Markkula R, Kalso E. Glucose tolerance in fibromyalgia. Medicine (Baltimore). 2021 Nov 19;100(46):e27803. doi: 10.1097/MD.0000000000027803. PMID 34797307
- [Derived] Zetterman T, Markkula R, Partanen JV, Miettinen T, Estlander AM, Kalso E. Muscle activity and acute stress in fibromyalgia. BMC Musculoskelet Disord. 2021 Feb 14;22(1):183. doi: 10.1186/s12891-021-04013-1. PMID 33583408